CLINICAL TRIAL: NCT04438330
Title: The Immunological Profile of Nickel Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Allergy Research Center, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-19080328
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-04

CONDITIONS: Nickel; Eczema; Nickel Sensitivity; Allergy; Inflammatory Response
Keywords: Patch test; metal allergy
MeSH Terms: conditions — Eczema; Hypersensitivity | interventions — nickel sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nickel allergic individuals (Experimental): Nickel sulfate hexahydrate in petrolatum. Exposed in a patch test dose-range with a max concentration of 5% nickel sulfate hexahydrate
  Interventions: Other: Nickel sulfate hexahydrate
- non-nickel allergic individuals (Active Comparator): Nickel sulfate hexahydrate in petrolatum. Exposed in a patch test dose-range with a max concentration of 5% nickel sulfate hexahydrate
  Interventions: Other: Nickel sulfate hexahydrate

INTERVENTIONS:
Other: Nickel sulfate hexahydrate — Patch test

SUMMARY:
A dose-response study on the immune phenotype of allergic nickel dermatitis on a previously exposed skin area.

DETAILED DESCRIPTION:
Clinically controlled study comprising 15 people with known nickel allergy and 15 healthy persons as control group. At the Department of Allergy and Dermatology, Gentofte Hospital, test participants will be exposed to nickel sulfate in a patch test on their back, which will create an eczema reaction in people with nickel allergy and induce skin resident T-cells. The resident T-cells will enhance further exposure. The eczema is healed over 3-4 weeks, after which the same areas are again exposed to nickel sulfate at different concentrations in a patch test. Skin biopsies of the exposed areas are taken and the immune phenotype is analyzed trough Nanostring RNA technologies of around 600 immunerelated genes.

ELIGIBILITY:
inclusion criteria

* Must be able to understand the written and oral participant information in Danish.
* Previously proven nick allergy by patch testing within the last 5 years, for the nickel allergic test participants.

exclusion criteria

* Pregnancy and / or breastfeeding.
* Systemic immunomodulatory treatments within the last 14 days.
* Local treatments of selected skin areas, such as applying hormone cream within the last two weeks or applying cream / lotion within 24 hours up to sample collection.
* Allergy to local anesthesia.
* Exposed to solar or sunlight on the back within 21 days.
* History of inflammatory skin diseases, asthma, Diabetes Mellitus, hives or arthritis (exclusion criteria only for participation in the healthy control group).
* Participation in another scientific experiment within the last 4 weeks. risks,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
mRNA Nanostring screening | 1 month
  Screening of 600 immune-related genes

SECONDARY OUTCOMES:
Protein verification | 2 month
  verification of differentially regulated mRNA at a protein level.

OTHER OUTCOMES:
Allergic response | 1 day
  Clinical evaluation of allergic response to a dose-range

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne D Johansen, Proff., Study Director — National Allergy Research Center, Denmark
Locations (1):
- National Allergy Research Center, Hellerup, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No